CLINICAL TRIAL: NCT02080689
Title: PROspective Study of the IMPACT of Decipher™ Prostate Cancer Classifier on Physician and Patient Treatment Consideration and Decisions Following Radical Prostatectomy [PRO-IMPACT]
Brief Title: Prospective Clinical Utility Study to Assess the Impact of Decipher on Treatment Decisions After Surgery
Acronym: PRO-IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GenomeDx Biosciences Corp (Industry)
Collaborators: Society of Urologic Oncology (SUO) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CU 004
Record Dates: First submitted 2014-02-18; First posted 2014-03-06 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Salvage setting (Other): The clinical utility of Decipher will be evaluated for patients meeting the inclusion criteria in the salvage setting: post-RP with evidence of PSA rise or BCR (defined as PSA detectable and rising on 2 or more subsequent determinations)
  Interventions: Other: Decipher
- Adjuvant setting (Other): The clinical utility of Decipher will be evaluated for patients in the adjuvant setting: within 12 months after surgery (in the absence of detectable PSA rise of BCR)
  Interventions: Other: Decipher

INTERVENTIONS:
Other: Decipher

SUMMARY:
The influence of Decipher test on urologist and patient treatment plan choices immediately post RP and at the time of PSA rise or BCR

DETAILED DESCRIPTION:
This prospectively decision impact study will evaluate physicians and patient treatment plan choices before and after reviewing Decipher results for eligible patient cases. The clinical utility of Decipher will be evaluated for patients meeting the inclusion criteria at two time-points post-RP:

1. In the adjuvant setting: within 12 months after surgery (in the absence of detectable PSA rise of BCR)
2. In the salvage setting: post-RP with evidence of PSA rise or BCR (defined as PSA detectable and rising on 2 or more subsequent determinations)

A total of 150 patient cases, in each arm, will be prospectively selected from clinical sites. The study as a whole will enroll 300 patient cases.

As a condition of participation in the study, each clinical site must agree to provide a minimum of 10 patient cases.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological T3 stage of disease (i.e., EPE or SVI), or
2. Positive surgical margins, or
3. Detectable PSA, defined as PSA detectable and rising on 2 or more subsequent determinations

Exclusion Criteria:

1. For adjuvant setting patients: Metastatic Disease (M+) prior to surgery
2. For salvage setting patients: Metastatic Disease at PSA rise
3. Failure of PSA to nadir after surgery
4. Received any neo-adjuvant prostate cancer treatment before radical prostatectomy
5. Received any adjuvant chemotherapy
6. Required patient clinical data is not available for evaluation of eligibility criteria
7. For adjuvant setting patients, any treatment received after surgery
8. For salvage setting patients, lack of documented treatment or management recommendation on file
9. Tissue specimen is inadequate for sampling and analysis

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2014-05; Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Number of participants for which the Decipher test changes the urologist's and patient's treatment plan choices | 3 months

SECONDARY OUTCOMES:
Measure the number of participants for which treatment was Increased or decreased in the intensity. | 3 months
  This outcome will compare recommended treatment pre-Decipher to recommended treatment post-Decipher
The number of different treatment plans most influenced by Decipher as a measure of clinical utility | 12 months
Comparison of type of treatment plans between high risk and low risk patients | 6 months
  How many treatment plans are similar for those considered at high versus low risk by Decipher test
Account for the number of specific treatment assignments that correlated with a change in treatment recommendation | 12 months
Frequency of follow visits as a measure of reproducibility | 12 months
  The extent to which the Decipher test results influence urologist recommendations on frequency of follow-up for patients
Measure the urologist's and patient's Level of confidence in their selected treatment plan through the use of a share decision making tool | 3 months
Assess the number of physicians that assigned the same treatment treatment recommendations for patient of the same pathological profile as a measure of concordance | 12 months
A measure of the patient's quality of life (QOL) as a measure of Decipher's clinical utility for patients | 12 months
  The extent to which the Decipher test results affect patient comfort level with treatment decisions as based on QOL and treatment regret tools
Evaluate number of participants which show coherence to treatment decisions | 12 months
  For how many cases was the original selected treatment for a patient actually executed upon

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W Lin, MD, Principal Investigator — The Society of Urologic Oncology (SUO); John L Gore, MD, Principal Investigator — University of Washington
Locations (19):
- United States (19):
  - Alaska Urology Institute Alaska Clinical Research Center, Anchorage, Alaska
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Colorado, Denver Medical Campus, Aurora, Colorado
  - The Urology Center of Colorado, Denver, Colorado
  - Urological Research Network, Hialeah, Florida
  - Lakeland Regional Health Systems, Lakeland, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Spectrum Health Medical Group, Grand Rapids, Michigan
  - Delaware Valley Urology, LLC, Voorhees Township, New Jersey
  - Carolina Urology Partners, Gastonia, North Carolina
  - Lancaster Urology, Lancaster, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Huntsman Cancer Hospital, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Virginia Urology, Richmond, Virginia
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Nguyen PL, Gu X, Lipsitz SR, Choueiri TK, Choi WW, Lei Y, Hoffman KE, Hu JC. Cost implications of the rapid adoption of newer technologies for treating prostate cancer. J Clin Oncol. 2011 Apr 20;29(12):1517-24. doi: 10.1200/JCO.2010.31.1217. Epub 2011 Mar 14. PMID 21402604
- [Background] Swanson GP, Basler JW. Prognostic factors for failure after prostatectomy. J Cancer. 2010 Dec 7;2:1-19. PMID 21197260
- [Background] Silberstein JL, Vickers AJ, Power NE, Fine SW, Scardino PT, Eastham JA, Laudone VP. Reverse stage shift at a tertiary care center: escalating risk in men undergoing radical prostatectomy. Cancer. 2011 Nov 1;117(21):4855-60. doi: 10.1002/cncr.26132. Epub 2011 Apr 11. PMID 21484780
- [Background] Thompson IM, Tangen CM, Paradelo J, Lucia MS, Miller G, Troyer D, Messing E, Forman J, Chin J, Swanson G, Canby-Hagino E, Crawford ED. Adjuvant radiotherapy for pathological T3N0M0 prostate cancer significantly reduces risk of metastases and improves survival: long-term followup of a randomized clinical trial. J Urol. 2009 Mar;181(3):956-62. doi: 10.1016/j.juro.2008.11.032. Epub 2009 Jan 23. PMID 19167731
- [Background] Bolla M, van Poppel H, Tombal B, Vekemans K, Da Pozzo L, de Reijke TM, Verbaeys A, Bosset JF, van Velthoven R, Colombel M, van de Beek C, Verhagen P, van den Bergh A, Sternberg C, Gasser T, van Tienhoven G, Scalliet P, Haustermans K, Collette L; European Organisation for Research and Treatment of Cancer, Radiation Oncology and Genito-Urinary Groups. Postoperative radiotherapy after radical prostatectomy for high-risk prostate cancer: long-term results of a randomised controlled trial (EORTC trial 22911). Lancet. 2012 Dec 8;380(9858):2018-27. doi: 10.1016/S0140-6736(12)61253-7. Epub 2012 Oct 19. PMID 23084481
- [Background] Wiegel T, Bottke D, Steiner U, Siegmann A, Golz R, Storkel S, Willich N, Semjonow A, Souchon R, Stockle M, Rube C, Weissbach L, Althaus P, Rebmann U, Kalble T, Feldmann HJ, Wirth M, Hinke A, Hinkelbein W, Miller K. Phase III postoperative adjuvant radiotherapy after radical prostatectomy compared with radical prostatectomy alone in pT3 prostate cancer with postoperative undetectable prostate-specific antigen: ARO 96-02/AUO AP 09/95. J Clin Oncol. 2009 Jun 20;27(18):2924-30. doi: 10.1200/JCO.2008.18.9563. Epub 2009 May 11. PMID 19433689
- [Background] Zelefsky MJ, Eastham JA, Cronin AM, Fuks Z, Zhang Z, Yamada Y, Vickers A, Scardino PT. Metastasis after radical prostatectomy or external beam radiotherapy for patients with clinically localized prostate cancer: a comparison of clinical cohorts adjusted for case mix. J Clin Oncol. 2010 Mar 20;28(9):1508-13. doi: 10.1200/JCO.2009.22.2265. Epub 2010 Feb 16. PMID 20159826
- [Background] Thompson IM Jr, Tangen CM, Paradelo J, Lucia MS, Miller G, Troyer D, Messing E, Forman J, Chin J, Swanson G, Canby-Hagino E, Crawford ED. Adjuvant radiotherapy for pathologically advanced prostate cancer: a randomized clinical trial. JAMA. 2006 Nov 15;296(19):2329-35. doi: 10.1001/jama.296.19.2329. PMID 17105795
- [Background] Hoffman KE, Nguyen PL, Chen MH, Chen RC, Choueiri TK, Hu JC, Kuban DA, D'Amico AV. Recommendations for post-prostatectomy radiation therapy in the United States before and after the presentation of randomized trials. J Urol. 2011 Jan;185(1):116-20. doi: 10.1016/j.juro.2010.08.086. Epub 2010 Nov 12. PMID 21074194
- [Background] Moinpour CM, Hayden KA, Unger JM, Thompson IM Jr, Redman MW, Canby-Hagino ED, Higgins BA, Sullivan JW, Lemmon D, Breslin S, Crawford ED, Southwest Oncology Group. Health-related quality of life results in pathologic stage C prostate cancer from a Southwest Oncology Group trial comparing radical prostatectomy alone with radical prostatectomy plus radiation therapy. J Clin Oncol. 2008 Jan 1;26(1):112-20. doi: 10.1200/JCO.2006.10.4505. PMID 18165645
- [Background] Erho N, Crisan A, Vergara IA, Mitra AP, Ghadessi M, Buerki C, Bergstralh EJ, Kollmeyer T, Fink S, Haddad Z, Zimmermann B, Sierocinski T, Ballman KV, Triche TJ, Black PC, Karnes RJ, Klee G, Davicioni E, Jenkins RB. Discovery and validation of a prostate cancer genomic classifier that predicts early metastasis following radical prostatectomy. PLoS One. 2013 Jun 24;8(6):e66855. doi: 10.1371/journal.pone.0066855. Print 2013. PMID 23826159
- [Background] Karnes RJ, Bergstralh EJ, Davicioni E, Ghadessi M, Buerki C, Mitra AP, Crisan A, Erho N, Vergara IA, Lam LL, Carlson R, Thompson DJ, Haddad Z, Zimmermann B, Sierocinski T, Triche TJ, Kollmeyer T, Ballman KV, Black PC, Klee GG, Jenkins RB. Validation of a genomic classifier that predicts metastasis following radical prostatectomy in an at risk patient population. J Urol. 2013 Dec;190(6):2047-53. doi: 10.1016/j.juro.2013.06.017. Epub 2013 Jun 11. PMID 23770138
- [Background] Badani K, Thompson DJ, Buerki C, Davicioni E, Garrison J, Ghadessi M, Mitra AP, Wood PJ, Hornberger J. Impact of a genomic classifier of metastatic risk on postoperative treatment recommendations for prostate cancer patients: a report from the DECIDE study group. Oncotarget. 2013 Apr;4(4):600-9. doi: 10.18632/oncotarget.918. PMID 23592338
- See also: The Society of Urologic Oncology (SUO) — http://suonet.org/default.aspx